CLINICAL TRIAL: NCT06518031
Title: The Effects of Meditation on Stress and Fatigue in Intensive Care Nurses: A Randomized Controlled Trial
Brief Title: The Effects of Meditation on Stress and Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Songul Gungor, Phd Lecturer, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: OKUKAU
Record Dates: First submitted 2024-07-16; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Intensive Care Nurses
Keywords: Meditation; Stress; Fatigue; Intensive Care Nurses; Well-being
MeSH Terms: conditions — Fatigue | interventions — Meditation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation Group (Experimental): Meditation practices were administered by the meditation expert for 6 weeks, three times a week for 20 minutes each session, totaling 60 minutes per week
  Interventions: Other: meditation
- Control Group (No Intervention): The research data were collected using a Personal Information Form prepared by the researchers containing introductory information about the nurses, the Perceived Stress Scale for stress, and the Fatigue Severity Scale for fatigue.

INTERVENTIONS:
Other: meditation — meditation practices were administered by the meditation expert for 6 weeks, three times a week for 20 minutes each session, totaling 60 minutes per week
  Arms: Meditation Group

SUMMARY:
A randomized controlled trial was conducted with nurses practicing meditation for six weeks, compared to a control group with no intervention. Stress and fatigue levels were measured using validated scales at baseline and post-intervention.

DETAILED DESCRIPTION:
Participants in the intervention group underwent a meditation practice for 20 minutes, three times a week for six weeks. The meditation sessions were led by a meditation expert with 8 years of experience and conducted online via WhatsApp in a group setting. No intervention was given to the participants in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care nurses with at least 1 year of experience in the intensive care unit.
* Nurses without chronic obstructive pulmonary disease, heart failure, asthma, or other conditions that could hinder breathing exercises.
* Nurses without hearing and communication issues, psychiatric diagnoses (e.g., major depression).
* Nurses who have not attended meditation, yoga, or breathing exercise classes in the past six months.
* Nurses willing to participate in the study were included in the sample.

Exclusion Criteria:

* Nurses who do not attend at least one of the meditation sessions conducted by the meditation expert.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-19 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
STRESS LEVELS | after 6 weeks
  PERCEIVED STRESS SCALE
FATIGUE LEVELS | after 6 weeks
  FATIGUE SEVERITY SCALE

CONTACTS AND LOCATIONS:
Locations (1):
- Songül GÜNGÖR, Merkez, Osmani̇ye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Purpose and Scope:
  This IPD plan outlines how individual participant data from the study "The Effects of Meditation on Stress and Fatigue in Intensive Care Nurses" will be shared and utilized. The data will be made available for verification of the study's findings and for further analysis by relevant researchers and scientific communities.
  Data Protection and Privacy:
  Participant data will be stored in compliance with national and international regulations to protect confidentiality. Data will only be shared for research purposes, ensuring participant identities are protected.
  Data Sharing Procedures:
  Data will be provided upon request to researchers and relevant institutions seeking to verify study results. Use of the data will be subject to approval by relevant ethics committees and for purposes of data sharing.
  Analysis Procedures:
  Data will be analyzed according to pre-established protocols, and findings will be presented in scientific reports. The methodology of analysis and i